CLINICAL TRIAL: NCT03505619
Title: Evaluation of an Intervention Program Addressing Reablement Services in a Swedish Context (ASSIST 1.0) - A Protocol for a Feasibility Study
Brief Title: ASSIST 1.0 an Intervention Program Addressing Reablement Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Susanne Guidetti, Principal Investigator, PhD, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASSIST 1.0
Record Dates: First submitted 2018-01-22; First posted 2018-04-23 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Older Adults; Participation
Keywords: home care service; reablement service; rehabilitation

STUDY DESIGN:
Intervention Model Description: A feasibility study with a pre-post-test design.
Who Masked: Participant, Care Provider
Masking Description: The older adults will be included if they fulfil the following inclusion criteria a) ≥65 years or older and live at home, b) home care has been granted and the user is deemed not to need home rehabilitation performed by rehabilitation staff, c) two or more identified challenges in everyday activities that can benefit from everyday rehabilitation, d) are able to understand and express themselves in Swedish. One or more of the reasons will result in exclusion from the study: have cognitive limitations that make reablement unappropriate, in need of care in institutional dwelling or are terminally ill ,the older adults have had home help services more than three years.
  When the older person in either the intervention or control group agrees to be involved in the study, they will be asked if they could consider involving a significant other.
  The home care providers delivering ASSIST 1.0 or the ordinary home care will be included consisting of 8-10 staff from each group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIST 1.0 (Experimental): A ten-week intervention program using a person-centred approach to support the older person to set up goals to perform daily activities that he/she wants or needs to do. The activity goals will target improvements in quality of life, physical health, mental well-being, and conditions for social community. The focus will be on supporting the older person's activities in everyday life that are considered meaningful for the individual. During the intervention, a specially designed application will send reminders and feedback related to the older adults' activity goals of doing their prioritized everyday activities both to the older adults and to the home care providers via mobile phones, tablet etc. The home care providers will participate in coaching sessions supporting the intervention held by the team of researchers.
  Interventions: Behavioral: ASSIST 1.0
- Ordinary home care services (No Intervention): The home care providers in the control group (CG) will provide services as usual to older adults participating in the control group. They will however, identify potential older persons to participate in the control group according to the same procedure and criteria as the intervention group.

INTERVENTIONS:
Behavioral: ASSIST 1.0 — 10 weeks intervention applying a person-centred approach by using goal setting and smart products.
  Arms: ASSIST 1.0

SUMMARY:
Reablement holds a potential to become a new rehabilitation model and has been implemented in some western countries including Norway and Denmark. At present, there is a lack of scientific evidence for the effectiveness of reablement and lack of an explicit theoretical underpinning, leading to a gap in knowledge. Trends show, however, that reablement is beneficial for the person and their significant others, increasing quality of life. There is a need for further investigation of the effects among community-dwelling adults in terms of clinical and economic outcomes. This research project will investigate the effectiveness of reablement including smart products (digitally based) (ASSIST) to facilitate and manage reablement services in home-dwelling adults compared with standard home help services in terms of daily activities, physical functioning, health-related quality of life, coping, mental health, use of health care services, and costs.

Methods and analysis: This feasibility study will evaluate the perceived value and acceptability of ASSIST 1.0 intervention program as the fidelity, reach and dose, and potential outcomes by using a pre-post test design involving an intervention group and a control group (n=30). All participants will be living at home and with a need of home care services. Qualitative interviews among home care providers delivering ASSIST and older adults and their significant others receiving the intervention will be conducted to explore aspects affecting the intervention.

Ethics and dissemination: The results will form the base for refinement of the "ASSIST" program and planning of a large-scale randomized, controlled trial investigating the effect of the program on quality of life as physical health, mental well-being, conditions for social community when focusing on supporting the older person's to meaningful everyday life. Dissemination will include peer-reviewed publications and presentations at national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years or older and live at home,
* home care has been granted and the user is deemed not to need home rehabilitation performed by rehabilitation staff,
* two or more identified challenges in everyday activities that can benefit from everyday rehabilitation,
* are able to understand and express themselves in Swedish.

Exclusion Criteria:

* have cognitive limitations that make reablement unappropriate,
* in need of care in institutional dwelling or are terminally ill ,
* the older adults have had home help services more than three years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) | Change between baseline and 8 to 10 weeks post baseline.
  Measuring the older adults' self-perception of activity performance and satisfaction within the areas of self care, productivity and leisure, measured on a 1-10 scale, where 10 represents most satsified and highest performance ranking.

SECONDARY OUTCOMES:
Change in Barthel Index | Change between baseline and 8 to 10 weeks post baseline.
  The Barthel Index (BI) will be administered at inclusion and post baseline will used in the present study to determine stroke severity, where scores of < 15 represented a severe stroke, 15-49 a moderate stroke, and 50-100 a mild stroke.
Frenchay Activity Index (FAI) | Change between baseline and 8 to 10 weeks post baseline.
  The FAI consist of 15 items, the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months, and ranges from 0 (inactive) to 45 (very active).
The Swedish version of the General Self -Efficacy Scale)(GSE) | Change between baseline and 8 to 10 weeks post baseline.
  Measure the perceived belief in one's ability in different situations. The GSE scale consists of ten statements such as "I can solve most problems if I invest the necessary effort." Possible responses are scored 1-4, where 1 represents "Not at all true", 2 "Hardly true", 3 "Moderately true" and 4 "Exactly true". This gives a total score ranging from 10-40; higher scores indicate a greater sense of general self-efficacy. The GSE has been translated into Swedish and has been demonstrated to be valid.
EQ5-D | Change between baseline and 8 to 10 weeks post baseline.
  EQ5-D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale.
Hospital Anxiety and Depression Scale (HAD) | Change between baseline and 8 to 10 weeks post baseline.
  The HADS is a screening instrument, which comprises Anxiety and Depression subscales, each with seven items and total scores ranging from 0-21. Higher scores indicate lower mood, i.e., more anxiety or depressive symptoms respectively. The recommended cut-offs for both subscales in people with stroke is ≥4
Mental Health Continuum -short form, Swedish version (MHC-SF) | Change between baseline and 8 to 10 weeks post baseline.
  Measure emotional well-being, social well-being and psychological well-being.
Reintegration of Normal Living Index- (RNL) | Change between baseline and 8 to 10 weeks post baseline.
  The RNLI index is made up of 11 declarative statements (e.g. I move around my living quarters as I feel necessary), including the following domains: indoor, community, and distance mobility; self-care; daily activity (work and school); recreational and social activities;; family role(s); personal relationships; presentation of self to others and general coping skills. The first 8 items represent 'daily functioning' and the remaining 3 items represent 'perception of self'.Each domain is accompanied by a visual analogue scale (VAS) (0 to 10 cm). The VAS is anchored by the statements "does not describe my situation" (1 or minimal integration) and "fully describes my situation" (10 or complete integration). Individual item scores are summed to provide a total score out of 110 points that is proportionally converted to create a score out of 100.
Change in Sense of Coherence | Change between baseline and 8 to 10 weeks post baseline.
  Short form measure on one's sense of health.
Change in Katz ADL extended scale | Change between baseline and 8 to 10 weeks post baseline.
  The Katz Extended Scale (KE) will be used to assess self-reported need of assistance (yes/no) in six personal ADL (PADL) and four instrumental ADL (IADL) both pre- and post-stroke.

OTHER OUTCOMES:
Creative Climate Questionnaire (CCQ) | Change between baseline and 8 to 10 weeks post baseline.
  Will measure the home care providers perceptions of organizational climate
QPS Nordic | Change between baseline and 8 to 10 weeks post baseline.
  Assessment for the home care providers psychological and social factors in the work place
Life Satisfaction Questionnaire (LiSat -11) | Change between baseline and 8 to 10 weeks post baseline.
  To assess life satisfaction the Life Satisfaction Scale (LiSat-11) (22) will be used. The LiSat-11contains 11 items about overall and domain-specific life satisfaction, self-rated on an ordinal scale ranging from 6 (very satisfactory) to 1 (very dissatisfactory). One global question assessing the participants' overall satisfaction with life.
Caregiver Burden Scale | Change between baseline and 8 to 10 weeks post baseline.
  The Caregiver Burden Scale (CBS) will be used to assess caregiver burden. The CBS consists of 22 items for different types of subjective caregiver burden, covering areas of the caregiver's health, feelings of psychological wellbeing, relations, social network, physical workload, and environmental aspects. The items are scored on a scale from 1 to 4 and the higher the score the greater the burden. The scale has been shown to have good construct validity and test-retest stability.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Borell, professor, Study Chair — Karolinska Institutet
Locations (1):
- Stockholms Äldre förvaltning, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Assander S, Bergstrom A, Eriksson C, Meijer S, Guidetti S. ASSIST: a reablement program for older adults in Sweden - a feasibility study. BMC Geriatr. 2022 Jul 26;22(1):618. doi: 10.1186/s12877-022-03185-2. PMID 35879678
- [Derived] Bergstrom A, Borell L, Meijer S, Guidetti S. Evaluation of an intervention addressing a reablement programme for older, community-dwelling persons in Sweden (ASSIST 1.0): a protocol for a feasibility study. BMJ Open. 2019 Jul 24;9(7):e025870. doi: 10.1136/bmjopen-2018-025870. PMID 31345964